CLINICAL TRIAL: NCT01370915
Title: Perioperative Administration of Pregabalin for Pain After Septoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Hun Jong Dhong, Professor, Department of Otorhinolaryngology-H&N surgery, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2010-06-012
Record Dates: First submitted 2011-04-20; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Deviated Nasal Septum
Keywords: postoperative pain, nasal septum surgery, pregabalin
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Patients receive oral placebo 150 mg 1hour prior to septal surgery, and 12 hours later
  Interventions: Drug: Pregabalin (Lyrica)
- Placebo (Placebo Comparator): Patients receive oral Placebo(Vitamin complex) 150 mg 1 hour before septal surgery, and 12 hours later
  Interventions: Drug: Vitamin complex (placebo)

INTERVENTIONS:
Drug: Pregabalin (Lyrica) — Patients receive oral Pregabalin 150 mg 1 hour before septal surgery, and 12 hours later
  Other Names: pregabalin
  Arms: Pregabalin
Drug: Vitamin complex (placebo) — Patients receive oral Placebo(Vitamin complex) 150 mg 1 hour before septal surgery, and 12 hours later
  Other Names: placebo, vitamin complex
  Arms: Placebo

SUMMARY:
Pregabalin is used for the treatment of neuropathic pain and has shown analgesic efficacy in postoperative pain. The aim of this randomized, double-blinded, placebo-controlled trial was to investigate the efficacy and safety of pregabalin for reducing postoperative pain in patients after septoplasty. Persons who scheduled for elective septoplasty under general anesthesia were randomly assigned to groups that received either pregabalin (150 mg twice) or placebo, one hour before surgery and 12 hours after the initial dose. Assessments of pain (verbal numerical rating scale) and side effects were performed at one, six, 12, and 24 hours postoperatively.

DETAILED DESCRIPTION:
Pregabalin is used for the treatment of neuropathic pain and has shown analgesic efficacy in postoperative pain. The aim of this randomized, double-blinded, placebo-controlled trial was to investigate the efficacy and safety of pregabalin for reducing postoperative pain in patients after septoplasty. Patients will be randomly assigned to one of two groups to receive either pregabalin (Lyrica®, Pfizer, Inc.) or placebo (vitamin complex). According to their assigned study group, patients received either pregabalin (75 mg) or placebo twice, one hour before surgery and 12 hours after the initial dose. The assessment of pain and side effects, such as nausea and vomiting, headache, dizziness, sedation, and blurred vision, were made at one, six, 12, and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 ≥ and ≤ 65 years
* Patients with nasal packing after septoplasty

Exclusion Criteria:

* previous septal surgery history
* postoperative complications including septal hematoma, bleeding ets.
* Current therapy with pregabalin, gabapentin, or any opioid
* Renal insufficiency
* History of seizure disorder

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Pain score (Verbal numerical rating scale, VNRS and Visual Analogue Scale, VAS) | postoperative 24 hrs

SECONDARY OUTCOMES:
The number of patients with side effects including Nausea and vomiting, sedation, headache, dizziness | postoperative 1, 6, 12, 24 hours
The number of patients who required additional analgesics during admission | postoperative 1,6,12,24 hour
Pain score (Verbal numerical rating scale, VNRS and Visual Analogue Scale, VAS) | postoperative 1, 6, 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hun Jong Dhong, MD, PhD, Principal Investigator — Samsung Medical Center, Department of Otorhinolaryngoloty
Locations (1):
- Department of Otorhinolaryngology H&N surgery, Sungkyunkwan University College of Medicine, Samsung Seoul Hospital, Seoul, South Korea